CLINICAL TRIAL: NCT01095250
Title: A 28-week Multicenter, Randomized, Double-masked, Placebo Controlled, Dose-ranging Phase III Study to Assess AIN457 Versus Placebo in Inducing and Maintaining Uveitis Suppression in Adults With Active, Non-infectious, Intermediate, Posterior or Panuveitis Requiring Immunosuppression (INSURE Study)
Brief Title: Safety and Efficacy of AIN457 in Patients With Active Non-infectious Uveitis
Acronym: INSURE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated: Study in Behcet's disease with mostly active uveitis did not meet its primary endpoint.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457C2302; 2009-014834-22
Record Dates: First submitted 2010-03-25; First posted 2010-03-30 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Uveitis
Keywords: Active uveitis; intermediate uveitis; panuveitis; posterior uveitis; uveitis
MeSH Terms: conditions — Uveitis; Uveitis, Intermediate; Panuveitis; Uveitis, Posterior | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- AIN457 300mg s.c every 2 weeks (Experimental): AIN457 300 mg s.c. at baseline, Week 1 and Week 2, then every 2 weeks.
  Interventions: Drug: AIN457
- AIN457 300mg s.c. every 4 weeks (Experimental): AIN457 300 mg s.c. at baseline and Week 2, then every 4 weeks.
  Interventions: Drug: AIN457
- AIN457 150mg s.c every 4 weeks (Experimental): AIN457 150 mg s.c. at baseline and Week 2, then every 4 weeks
  Interventions: Drug: AIN457
- Placebo s.c every 2 weeks (Placebo Comparator): Placebo s.c at baseline, Week 1 and Week 2, then every 2 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AIN457
  Arms: AIN457 300mg s.c every 2 weeks
Drug: AIN457
  Arms: AIN457 150mg s.c every 4 weeks
Drug: AIN457
  Arms: AIN457 300mg s.c. every 4 weeks
Drug: Placebo
  Arms: Placebo s.c every 2 weeks

SUMMARY:
This study will assess the safety and efficacy of AIN457 as adjunctive therapy for the treatment of intermediate uveitis, posterior uveitis, or panuveitis requiring systemic immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥18 years of age. Where relevant, parents will also sign the informed consent according to local laws and regulations
* Patients with diagnosis of chronic non-infectious intermediate uveitis, posterior uveitis or panuveitis in at least one eye
* Evidence of active intermediate, posterior or panuveitis (grade ≥ 2+ vitreous haze with or without the presence of anterior chamber cells) at screening and baseline in at least one eye
* Requirement for any of the following immunosuppressive therapies for the treatment or prevention of uveitis:
* Prednisone or equivalent ≥10 mg daily at any time within the past 3 months.
* ≥1 periocular injection or ≥1 intravitreal corticosteroid injection (e.g. triamcinolone) in the study eye within the past 6 months (the last injection must not have been given 6 weeks prior to screening).
* Treatment with either cyclosporine, tacrolimus, azathioprine, mycophenolate mofetil, mycophenolic acid, methotrexate at any time within the past 3 months (Patients treated with chlorambucil or cyclophosphamide within the past 5 years are ineligible for the study).
* Patients not meeting the above specified criteria for immunosuppressive therapies are eligible for enrollment if they are intolerant to systemic immunosuppressive therapy as determined by the study investigator.
* Patient must be able to understand and communicate with the investigator and comply with the requirements of the study and must give a written, signed and dated informed consent before any study assessment is performed

Exclusion Criteria:

Ocular concomitant conditions/disease

* Patients receiving or that may require prednisone (or equivalent) ≥1.5 mg/kg/day for the treatment of their active uveitis
* Patients with a primary diagnosis of Behcet's disease, anterior uveitis or any intermediate uveitis, posterior uveitis or panuveitis in which the manifestation(s) of the active intraocular inflammatory disease may spontaneously resolve or that are not characterized by the presence of either anterior chamber cells or vitritis (vitreous cell and haze) such as the white dot retino-choroidopathies (i.e. Punctate inner choroidopathy (PIC), acute zonal occult outer retinopathy (AZOOR)
* Patients with infectious uveitis or uveitis of an underlying diagnosis that is uncertain and would reasonably include a disease for which immunosuppression would be contraindicated (e.g. ocular lymphoma)

Ocular treatments

* Treatment with intravitreal anti-VEGF agents administered to the study eye within 3 months prior to screening
* Treatment with fluocinolone acetonide implant in the study eye within the last 3 years, or dexamethasone intravitreal implant and any other investigational corticosteroid implants in the study eye within the last 6 months.
* Intraocular surgery or laser photocoagulation in the study eye within the last 6 weeks prior to screening except for a diagnostic vitreous or aqueous tap with a small-gauge needle
* Ocular disease that would interfere with ocular evaluations (e.g. corneal scarring, cataract, vitreous hemorrhage) or that in the opinion of the investigator would complicate the evaluation of the safety or efficacy of the study treatment (e.g. uncontrolled glaucoma, toxoplasma scar, macular scarring)
* Current use of or likely need for systemic medications known to be toxic to the lens, retina, or optic nerve (e.g., deferoxamine, chloroquine, ethambutol, etc.)

Systemic conditions or treatments

* Any previous treatment with AIN457
* Any systemic biologic therapy (e.g. interferon, infliximab, daclizumab, etanercept, or adalimumab) given intravenously or subcutaneously within 3 months prior to screening. No biologic therapy other than the investigational study treatment will be allowed during the course of the clinical trial
* Any prior treatment with systemic alkylating agents (cyclophosphamide, chlorambucil) within the past 5 years prior to screening
* Treatment with any live or live-attenuated vaccine (including vaccine for varicella-zoster or measles) within 2 months prior to screening. No treatment with live or live-attenuated vaccines will be allowed during the course of the clinical trial

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (34):
- United States (5):
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Cambridge, Massachusetts
  - Novartis Investigative Site, Slingerlands, New York
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Houston, Texas
- Canada (3):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, North York, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Cairo, Egypt
- Novartis Investigative Site, Nantes, France
- Germany (2):
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Göttingen
- Novartis Investigative Site, Budapest, Hungary
- Novartis Investigative Site, Ahmedabad, Gujarat, India
- Israel (4):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Japan (9):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Shimotsuka-gun, Tochigi
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Mitaka, Tokyo
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Switzerland (4):
  - Novartis Investigative Site, Lausanne, CHE
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lucerne
  - Novartis Investigative Site, Sankt Gallen
- Novartis Investigative Site, York, United Kingdom

REFERENCES:
- [Derived] Dick AD, Tugal-Tutkun I, Foster S, Zierhut M, Melissa Liew SH, Bezlyak V, Androudi S. Secukinumab in the treatment of noninfectious uveitis: results of three randomized, controlled clinical trials. Ophthalmology. 2013 Apr;120(4):777-87. doi: 10.1016/j.ophtha.2012.09.040. Epub 2013 Jan 3. PMID 23290985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Disposition of the 31 randomized patients is summarized in the table below. As a consequence of the early termination, few patients (N=31) were randomized into this study. Of these, 30 patients were discontinued due to administrative reasons (30 patients due to study termination and also one due to misrandomization). One patient withdrew consent.
Pre-assignment Details: As a consequence of the early termination, few patients (N=31) were randomized into this study. Of these, 30 patients were discontinued due to administrative reasons (30 patients due to study termination, including one due to misrandomization. One patient withdrew consent.
Groups:
- AIN457 300mg s.c Every 2 Weeks: AIN457 300 mg subcutaneously at baseline, Week 1 and Week 2, then every 2 weeks
- AIN457 300mg s.c. Every 4 Weeks: AIN457 300 mg subcutaneously at baseline and Week 2, then every 4 weeks.
- AIN457 150mg s.c Every 4 Weeks: AIN457 150 mg subcutaneously at baseline and Week 2, then every 4 weeks.
Period: Overall Study
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c. Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks
Started | 8 | 10 | 8 | 5
Completed | 0 | 0 | 0 | 0
Not Completed | 8 | 10 | 8 | 5
Not completed — administrative reasons | 8 | 10 | 7 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c. Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks | Total
Number analyzed (Participants) | 8 | 10 | 8 | 5 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.5 (21.13) | 46.9 (12.80) | 44.6 (15.99) | 50.6 (12.99) | 47.1 (15.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 2 | 3 | 15
  Male | 4 | 4 | 6 | 2 | 16
Region of Enrollment [Number; unit: Participants]
  Canada | 0 | 2 | 1 | 1 | 4
  Switzerland | 0 | 1 | 0 | 0 | 1
  Germany | 0 | 0 | 0 | 1 | 1
  France | 0 | 0 | 1 | 0 | 1
  Hungary | 1 | 1 | 0 | 0 | 2
  Israel | 0 | 2 | 1 | 0 | 3
  Japan | 4 | 3 | 4 | 2 | 13
  Singapore | 1 | 0 | 0 | 0 | 1
  United States | 2 | 1 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Vitreous Haze Grade in the Study Eye From Baseline to 28 Weeks or at Time of Rescue, if Earlier.
Description: No patients of Study CAIN457C2303 achieved the milestone of the primary endpoint in non-infectious uveitis patients with Behçet's disease. Study CAIN457C2302 (active uveitis study) was terminated to avoid continuing patients on a study with a low probability of success.Since patients did not reach the endpoint of analysis there can be no meaningful interpretation of data and data will be not provided.
Time Frame: baseline to 28 weeks
Population: The results of Study CAIN457C2303 did not meet the primary endpoint in non-infectious uveitis patients with Behçet's disease. Study CAIN457C2302 (active uveitis study) was terminated to avoid continuing patients on a study with a low probability of success.
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c. Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Proportion of Responders With no Recurrence of Active Intermediate, Posterior, or Panuveitis in the Study Eye at 28 Weeks
Description: as for outcome 1
Time Frame: baseline to 28 weeks
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c. Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Mean Change in Best Corrected Visual Acuity From Baseline to 28 Weeks
Description: as for outcome 1
Time Frame: baseline to 28 weeks
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c. Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Quality of Life/Patient Reported Outcome Assessments
Description: as for outcome 1
Time Frame: baseline to 28 weeks
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c. Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Mean Change in Vitreous Haze Grade and Anterior Chamber Cell Grade From Baseline to 28 Weeks
Description: as for outcome 1
Time Frame: baseline to 28 weeks
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c. Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Change in Immunosuppressive Medication Score From Baseline to Week 28
Description: as for outcome 1
Time Frame: baseline to 28 weeks
Arm/Group | AIN457 300mg s.c Every 2 Weeks | AIN457 300mg s.c. Every 4 Weeks | AIN457 150mg s.c Every 4 Weeks | Placebo s.c Every 2 Weeks
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: One patient in the placebo arm was a misrandomized patient and did not receive any treatment and is not included in the adverse events section.
Groups:
- AIN457 300mg Every 2 Weeks: AIN457 300 mg s.c. at baseline, Week 1 and Week 2, then every 2 weeks
- AIN457 300mg Every 4 Weeks: AIN457 300 mg subcutaneously at baseline and Week 2, then every 4 weeks.
- AIN457 150mg Every 4 Weeks: AIN457 150 mg s.c. at baseline and Week 2, then every 4 weeks
- Placebo Every 2 Weeks: Placebo s.c at baseline, Week 1 and Week 2, then every 2 weeks
Arm/Group | AIN457 300mg Every 2 Weeks | AIN457 300mg Every 4 Weeks | AIN457 150mg Every 4 Weeks | Placebo Every 2 Weeks
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/10 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 6/8 | 4/10 | 6/8 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300mg Every 2 Weeks (N=8) | AIN457 300mg Every 4 Weeks (N=10) | AIN457 150mg Every 4 Weeks (N=8) | Placebo Every 2 Weeks (N=4)
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300mg Every 2 Weeks (N=8) | AIN457 300mg Every 4 Weeks (N=10) | AIN457 150mg Every 4 Weeks (N=8) | Placebo Every 2 Weeks (N=4)
Blepharitis (Fellow eye) (Eye disorders) | 0 | 0 | 0 | 1
Blepharitis (Study eye) (Eye disorders) | 0 | 0 | 0 | 1
Cataract (Fellow eye) (Eye disorders) | 0 | 0 | 1 | 0
Cataract nuclear (Fellow eye) (Eye disorders) | 0 | 0 | 1 | 0
Cataract nuclear (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Glaucoma (Fellow eye) (Eye disorders) | 0 | 1 | 0 | 0
Lacrimation increased (Fellow eye) (Eye disorders) | 0 | 0 | 0 | 1
Lacrimation increased (Study eye) (Eye disorders) | 0 | 0 | 0 | 1
Ocular sarcoidosis (Fellow eye) (Eye disorders) | 0 | 0 | 1 | 0
Ocular sarcoidosis (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Puncture site haemorrhage (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Cataract traumatic (Fellow eye) (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Eye injury (Fellow eye) (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1
Intraocular pressure increased (Fellow eye) (Investigations) | 0 | 0 | 0 | 1
Intraocular pressure increased (Study eye) (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Study CAIN457C2302 was terminated to avoid continuing patients on a study with a low probability of success. Since patients did not reach the endpoint of analysis there can be no meaningful interpretation of data and data will be not provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.